CLINICAL TRIAL: NCT06706258
Title: Post-Cardiac Surgery Acute Kidney Injury Prevention by Administration of Proton Pump Inhibitor (P2 Trial): A Prospective Randomized Controlled Trial
Brief Title: Post-Cardiac Surgery Acute Kidney Injury Prevention by Administration of Proton Pump Inhibitor (P2 Trial)
Acronym: P2 AKI PPI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, yafen liang, M.D.; Professor; Chief, Division of Cardiovascular Anesthesiology; Vice Chair, Clinical Research, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSC-MS-24-1034
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; AKI; Cardiac Surgery; Cardiovascular Surgery; PPI; Proton Pump Inhibitors; Perioperative Medicine; Anesthesiology; Intensive Care Unit; ICU; Kidney
MeSH Terms: conditions — Acute Kidney Injury | interventions — Pantoprazole; Famotidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pantoprazole Group (Experimental): Pantoprazole (Protonix) will be given at 6 different timepoints:
  1. After anesthesia induction, before surgical incision.
  2. At chest closure. 3 & 4. Every 12 hrs in post operative day 1. 5 & 6. Every 12 hrs in post operative day 2.
  Interventions: Drug: Protonix (Pantoprazole) 40 mg q 12 hrs for 3 days
- Famotidine Group (Active Comparator): Famotidine (Pepcid) will be given at 6 different timepoints:
  1. After anesthesia induction, before surgical incision.
  2. At chest closure. 3 & 4. Every 12 hrs in post operative day 1. 5 & 6. Every 12 hrs in post operative day 2.
  Interventions: Drug: Pepcid (Famotidine) 20 mg q 12 hrs for 3 days

INTERVENTIONS:
Drug: Protonix (Pantoprazole) 40 mg q 12 hrs for 3 days — Administer 1st dose after anesthesia induction before surgical incision, 2nd dose at chest closure. Then, every 12 hrs for 2 more days.
  Arms: Pantoprazole Group
Drug: Pepcid (Famotidine) 20 mg q 12 hrs for 3 days — Administer 1st dose after anesthesia induction before surgical incision, 2nd dose at chest closure. Then, every 12 hrs for 2 more days.
  Arms: Famotidine Group

SUMMARY:
The central hypothesis of this research study is that perioperative administration of the proton pump inhibitor (PPI) pantoprazole could reduce the development of acute kidney injury (AKI) following cardiac surgery by activation molecular pathways for kidney protection. The investigators propose a single-center, randomized, controlled, single-blinded trial to determine whether perioperative intravenous administration of pantoprazole will reduce the incidence of AKI, some molecules that can be detected the urine, and major adverse kidney events (MAKE) at day 30 postoperatively, compared to famotidine after cardiac surgery. The specific aims of the study will be achieved by randomizing a group of 400 patients to receive pantoprazole (study) or famotidine (control) for 3 days perioperatively.

Our study population will include any adult patients (aged over 18 years) scheduled for cardiac surgery requiring a cardiopulmonary bypass machine.

DETAILED DESCRIPTION:
Each year more than 500,000 cardiac surgeries are performed in the USA alone. AKI is a common complication following cardiac surgery and is associated with poor patient outcome and increased health care cost. Therefore, there is an urgent need to identify medical interventions and treatments that prevent AKI or mitigate its severity when it occurs after cardiac surgery.

One of the main causes of AKI following cardiac surgery involves renal hypoperfusion/ischemia and reperfusion injury. Hypoxia inducible factors (HIFs) are key transcription factors responsible for tissue adaptation to low oxygen, which orchestrate the expression of a wide variety of genes including a set of microRNAs. MicroRNAs are endogenous single-stranded noncoding miRNAs of nucleotides that participate in physiological and pathological functions via regulating post-transcription of target genes. During ischemic injury, hypoxia upregulates endothelial MicroRNAs that have a potential in renal protection through vascular integrity and regeneration. Additionally, microRNAs exert protective effects via decreasing apoptosis and promoting tubular cell proliferation during ischemic AKI. Moreover, decreased serum levels of MicroRNAs are highly correlated with AKI severity in the intensive care unit (ICU) patients.

Our preliminary study identified ATP4A as the downstream target gene of MicroRNAs in the kidney. ATP4A (catalytic α subunit of H+/K+ ATPase) is located in intercalated cells in the distal tubules and cortical collecting ducts, which regulates urine acidification through secretion of hydrogen and reabsorption of potassium from urine. Proton pump inhibitors (PPIs) block the ATP hydrolysis of the H+/K+ ATPase via binding its active site of ATP4A and further enhance this endogenous kidney protection pathway. Despite robust animal model data, randomized controlled trial aiming to test the effectiveness of PPI in post-cardiac surgery AKI prevention is lacking. If proven to be effective, our studies could be easily implemented in clinical practice and serve as an effective treatment for perioperative AKI.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18-90).
* Scheduled for elective cardiac surgery with cardiopulmonary bypass.
* Moderate to high risk of developing AKI (Cleveland risk score equal to or higher than 3.

Exclusion Criteria:

* Patients with preoperative eGFR<30 ml/min/1.73 m2
* Dialysis dependence
* Emergency surgery
* Pregnancy.
* Nursing patient
* Patients with interstitial nephritis
* PPIs hypersensitivity
* Liver disease
* Vitamin B12 deficiency.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Acute Kidney Injury (AKI) | From enrollment to 7 days or until hospital discharge, if earlier.
  The investigators will calculate the incidence of acute kidney injury (AKI) within 7 days (or until hospital discharge if earlier) of cardiac surgery in patients receiving pantoprazole vs. famotidine.

SECONDARY OUTCOMES:
Urinary Kidney Injury Biomarkers Levels | From enrollment to 72 hours after ICU admission
  The investigators will measure the urinary kidney biomarker KIM-1 (kidney injury molecule-1) and neutrophil gelatinase-associated lipocalin (NGAL) levels at the different time points of urine sample collection (baseline, chest closure, and 8, 24, 48 and 72 hrs after ICU admission)
Major Adverse Kidney Events (MAKE) | From enrollment to 30 days after cardiac surgery
  The investigators will follow up on patients enrolled in the study and ask about patient demise, necessity of dialysis of any type, hospitalizations due to renal problems, or sustained kidney dysfunction after 30 days of enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Yafen Liang, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Texas Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared upon request by the journal.
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be available and uploaded on clinicaltrials.gov website when it is due.
Access Criteria: Accesible through the clinicaltrials.gov website.
URL: https://register.clinicaltrials.gov/